CLINICAL TRIAL: NCT03156543
Title: Evaluation of a Microcurrent Dressing for Prophylaxis Against Perioperative Prosthetic Joint Infection
Brief Title: Microcurrent Dressing to Treat Infections, Before, During and After Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Arthrex, Inc. (Industry)
Responsible Party: Principal Investigator, Bruce Miller, MD-Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HUM00109957
Record Dates: First submitted 2017-05-08; First posted 2017-05-17 (Actual); Results first posted 2020-10-09 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-09

CONDITIONS: Shoulder Arthropathy Associated With Other Conditions; Shoulder Arthritis; Shoulder Osteoarthritis; Shoulder Pain
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group A (Experimental): This group will have the jumpstart dressing pre-operatively and a standard dressing post operatively.
  Interventions: Device: Jumpstart Dressing; Other: Standard Dressing
- Group B (Experimental): This group will have the jumpstart dressing pre-operatively and a jumpstart dressing post operatively.
  Interventions: Device: Jumpstart Dressing

INTERVENTIONS:
Device: Jumpstart Dressing — JumpStart™ is a wireless, advanced microcurrent generating, dressing used for the management of surgical incision sites. Microcell batteries made of silver and zinc, generate an electrical current when activated by conductive fluids, such as saline, hydrogel or wound exudate. These microcells create low voltage electrical fields to stimulate the surrounding area and to provide antimicrobial protection to assist with wound healing. JumpStart has demonstrated superior broad spectrum bactericidal activity of a wound dressing against antibiotic-resistant strains of wound isolates within 24 hours.
  It will be applied pre-op in all patients and post operatively in group B
Other: Standard Dressing — This is a standard of care bandage that will be placed on participants in group A post operatively
  Other Names: Gauze
  Arms: Group A

SUMMARY:
Deep periprosthetic infection following total joint arthroplasty is a major complication. Although it only occurs in a small percentage of patients (~1%), it results in substantial morbidity and a decline in functional outcome. A two stage revision and exchange is commonly required in order to clear the infection and provide the best opportunity for prosthetic replantation. Following removal of the infected components, a minimum course of six weeks of parenteral antibiotics is given and resolution of the infection confirmed through the ESR, CRP, and repeated aspiration of the joint. In most instances a temporary spacer of antibiotic-loaded cement is inserted at the first stage and removed at the second operation.

Propionibacterium Acnes is a gram-positive, non-spore-forming, anaerobic bacillus found in lipid-rich areas, including hair follicles, sebaceous glands, and moist areas of the shoulder and axilla. Because of its low virulence, infections caused by P. acnes typically have a low-grade, indolent course, with shoulder pain often the only presenting symptoms after prosthetic replacement. P. acnes is particularly challenging to both diagnose and to eradicate, and is a substantial source of morbidity with shoulder arthroplasty.

JumpStart™ is a wireless, advanced microcurrent generating, dressing used for the management of surgical incision sites. Microcell batteries made of silver and zinc, generate an electrical current when activated by conductive fluids, such as saline, hydrogel or wound exudate. These microcells create low voltage electrical fields to stimulate the surrounding area and to provide antimicrobial protection to assist with wound healing. JumpStart has demonstrated superior broad spectrum bactericidal activity of a wound dressing against antibiotic-resistant strains of wound isolates within 24 hours.

The use of JumpStart as a prophylactic preoperative dressing to alter the skin flora and thereby decrease the risk of prosthetic infection has not been investigated to-date. Given the morbidity of a prosthetic infection, this would be a remarkably valuable intervention for any joint replacement procedure.

ELIGIBILITY:
Inclusion Criteria:

* Limited to total or reverse shoulder arthroplasty
* All patients 18 years of age and older

Exclusion Criteria:

* Under the age of 18
* Revision shoulder arthroplasty patients
* Sensitivity or allergy to sliver or zinc or latex

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-04-19 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Jumpstart Dressing Pre-Operatively Only: This group will have the jumpstart dressing pre-operatively and a standard dressing post operatively.
  Jumpstart Dressing: JumpStart™ is a wireless, advanced microcurrent generating, dressing used for the management of surgical incision sites. Microcell batteries made of silver and zinc, generate an electrical current when activated by conductive fluids, such as saline, hydrogel or wound exudate. These microcells create low voltage electrical fields to stimulate the surrounding area and to provide antimicrobial protection to assist with wound healing. JumpStart has demonstrated superior broad spectrum bactericidal activity of a wound dressing against antibiotic-resistant strains of wound isolates within 24 hours.
  It will be applied pre-op in all patients and post operatively in group B
  Standard Dressing: This is a standard of care bandage that will be placed on participants in group A post operatively
- Jumpstart Dressing Pre and Post-Operatively: This group will have the jumpstart dressing pre-operatively and a jumpstart dressing post operatively.
  Jumpstart Dressing: JumpStart™ is a wireless, advanced microcurrent generating, dressing used for the management of surgical incision sites. Microcell batteries made of silver and zinc, generate an electrical current when activated by conductive fluids, such as saline, hydrogel or wound exudate. These microcells create low voltage electrical fields to stimulate the surrounding area and to provide antimicrobial protection to assist with wound healing. JumpStart has demonstrated superior broad spectrum bactericidal activity of a wound dressing against antibiotic-resistant strains of wound isolates within 24 hours.
  It will be applied pre-op in all patients and post operatively in group B
Period: Overall Study
Arm/Group | Jumpstart Dressing Pre-Operatively Only | Jumpstart Dressing Pre and Post-Operatively
Started | 9 | 23
Completed | 8 | 23
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Jumpstart Dressing Pre-Operatively Only | Jumpstart Dressing Pre and Post-Operatively | Total
Number analyzed (Participants) | 9 | 23 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.78 (7.54) | 59.64 (15.92) | 62.29 (14.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 6 | 18 | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 9 | 23 | 32

OUTCOME MEASURES:

1. Primary Outcome: Measurement of Change in Cutibacterium Acnes
Description: All topical and deep tissue specimens were planned to be cultured for Propionibacterium Acnes. The type and number of colony forming units (CFU) will be recorded. Propionibacterium was renamed during the course of the trial, so the actual bacteria culture was Cutibacterium.
  Swabs for topical bacteria collections were taken 48 hours apart; biopsies to check on bacterial depth were taken at time of surgery.
  Bacteria CFU counts were classified into 5 categories: None, Minimal, (1-5 colonies) Few, (6-15 colonies) Moderate (16-99 colonies) and Numerous (100 or greater).
  Participants are categorized by their initial count categories and their change (expressed as reduction, no change, or increase) in CFU count (categorized) as measured by skin swabs; Biopsy count category discrepancies from time of surgery swab are only shown if they were a more than 1 category difference.
Time Frame: 2 days pre-operatively and at the time of surgery
Population: Data analyzed only for participants who had both measurements
Measure: Count of Participants; unit: Participants
Arm/Group | Jumpstart Dressing Pre-Operatively Only | Jumpstart Dressing Pre and Post-Operatively
Number analyzed (Participants) | 9 | 22
Participants
  No Bacteria at Start; No change | 3 | 8
  Minimal Start; Decrease | 3 | 2
  Minimal Start; No change | 1 | 2
  Few Start; Decrease | 0 | 1
  Few Start; No change | 0 | 1
  Moderate Start; Decrease | 1 | 3
  Moderate Start; Increase | 0 | 1
  Numerous Start; Decrease | 0 | 1
  Numerous Start; No change | 0 | 2
  Few start; no change; 2 level increase biopsy only | 0 | 1
  Moderate Start; 3 level decrease; no change biopsy | 1 | 0
Statistical Analysis 1: Comparison: Jumpstart Dressing Pre-Operatively Only vs Jumpstart Dressing Pre and Post-Operatively; Analysis was based on the participants who were positive for C. acnes; Test type: Superiority; p = 0.004, Fisher Exact

2. Secondary Outcome: Cosmesis and Apposition
Description: Investigator determined from a small number of collected images that because of the number of arthroscopies rather than arthroplasties performed, the surgical wound was not large enough to evaluate the wound healing effect of dressings. Photo collection was discontinued and that data was not analyzed
Time Frame: At 7 days and then again 10-14 days postoperatively
Population: The original Principal Investigator had determined from a small number images that photos did not demonstrate sufficient differentiation to evaluate effect of dressings. The co-investigator who became the Principal Investigator neither resumed photo collection, nor analyzed those taken.
Arm/Group | Jumpstart Dressing Pre-Operatively Only | Jumpstart Dressing Pre and Post-Operatively
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 9 - 12 days from baseline to after surgery appointment (based on standard after-surgery appointment)
Arm/Group | Jumpstart Dressing Pre-Operatively Only | Jumpstart Dressing Pre and Post-Operatively
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/23
Other Adverse Events (participants affected / at risk) | 0/9 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2018-01-05): https://cdn.clinicaltrials.gov/large-docs/43/NCT03156543/Prot_000.pdf